CLINICAL TRIAL: NCT07027787
Title: Effect of Incentive Training on Hand Dexterity Skills in Male Stroke Patients: A Randomized Controlled Trial
Brief Title: Incentive Training Role in Treatment of Hand Dexterity in Patients With Stroke
Acronym: HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Collaborators: Princess Nourah Bint Abdulrahman University (Other); Keele University (Other); Cairo University (Other); Queen Margaret University (Other); Delta University for Science and Technology (Other); Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Omar Mohamed Kamel, researcher, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hand dexterity
Record Dates: First submitted 2025-06-16; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Stroke
Keywords: Incentive training; Attention; Hand dexterity; stroke
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Physical Therapy for Hand Dexterity in Stroke Patients (Active Comparator): Standard physical therapy program for stroke patients targeting hand dexterity. Conducted 3 times/week for 8 weeks (60 min/session), exercises included wrist and forearm movements, object manipulation, ball gripping, and putty-based hand strengthening.
  Interventions: Behavioral: Standard Physical Therapy for Hand Dexterity in Stroke Patients
- Rehacom Attention Training + Physical Therapy (Active Comparator): Combined intervention: 30 minutes of computerized attention training using the Rehacom system, followed by 30 minutes of standard hand dexterity physical therapy. Conducted 3 times/week for 8 weeks. Rehacom provided task-based cognitive training with visual, auditory, and performance feedback in a controlled lab setting.
  Interventions: Behavioral: Rehacom Attention Training + Physical Therapy

INTERVENTIONS:
Behavioral: Standard Physical Therapy for Hand Dexterity in Stroke Patients — Standard physical therapy program for stroke patients targeting hand dexterity. Conducted 3 times/week for 8 weeks (60 min/session), exercises included wrist and forearm movements, object manipulation, ball gripping, and putty-based hand strengthening.
  Arms: Standard Physical Therapy for Hand Dexterity in Stroke Patients
Behavioral: Rehacom Attention Training + Physical Therapy — Combined intervention: 30 minutes of computerized attention training using the Rehacom system, followed by 30 minutes of standard hand dexterity physical therapy. Conducted 3 times/week for 8 weeks. Rehacom provided task-based cognitive training with visual, auditory, and performance feedback in a controlled lab setting.
  Arms: Rehacom Attention Training + Physical Therapy

SUMMARY:
Attention and hand dexterity are interdependent, with deficits in one often worsening the other. Post-stroke, reduced attention impairs hand dexterity, hindering daily activities, while poor hand function further limits attentional focus. Despite progress in rehabilitation, strategies addressing both remain limited. Purpose: This study explored the impact of incentive-based attention training on hand dexterity in stroke patients.

DETAILED DESCRIPTION:
Forty male patients with hemorrhagic infarction stroke, aged 45-60 years, were randomized into two equal groups. The control group (Group A, n=20) underwent hand dexterity exercises for 60 minutes per session, while the intervention group (Group B, n=20) received a combination of 30 minutes of hand dexterity exercises and 30 minutes of attention training using the Rehacom system. Both groups completed three training sessions per week for eight weeks (24 sessions). Outcomes were assessed pre- and post-training using the Mindful Attention Awareness Scale (MAAS), Hand Grip Dynamometer, Rehacom system, and Purdue Pegboard Test (PPBT).

ELIGIBILITY:
Inclusion Criteria:

1. ) Male patients diagnosed with chronic hemorrhagic infarction stroke
2. ) Stroke diagnosis confirmed through CT or MRI scans
3. ) Referred by a neurologist or neurosurgeon
4. ) Right-handed
5. ) Aged between 45 and 60 years
6. ) Stroke duration ranging from 6 months to 1 year
7. ) Mini-Mental State Examination (MMSE) score of 24 or higher
8. ) Montreal Cognitive Assessment (MoCA) score above 21, indicating no significant cognitive impairment
9. ) Mild spasticity (Grade 1 or 1+ on the Modified Ashworth Scale)
10. ) Brunnstrom's Stage 4 or 5 of recovery

Exclusion Criteria:

1. ) Unstable medical conditions (e.g., diabetes mellitus or hypertension)
2. ) Language deficits that could impair cooperation
3. ) Blindness or deafness
4. ) Severe cognitive impairments affecting task performance
5. ) Presence of brain tumors

Ages: 45 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Hand dexterity assessment using the Purdue Pegboard Test (PPBT) | 8 Weeks
  The Purdue Pegboard Test (PPBT) is a timed neuropsychological assessment used to evaluate fine motor skills, finger dexterity, and bimanual coordination by measuring how quickly a person can place small pegs into holes using one or both hands.
Hand grip dynamometer (JAMAR) | 8 weeks
  The JAMAR hand dynamometer is a reliable and widely used tool for measuring grip strength, featuring a peak-hold needle and adjustable handle settings to accommodate different hand sizes and ensure consistent, accurate readings.

SECONDARY OUTCOMES:
Rehacom system | 8 Weeks
  The Rehacom system is a CE-certified, software-based cognitive rehabilitation tool that personalizes training and assessment in domains like attention, memory, and logic. This study utilizes its attention-concentration module to evaluate the cognitive performance of stroke patients through detailed reaction-time metrics and adaptive difficulty levels.
The Mindful Attention Awareness Scale (MAAS)( 6 is high 6 , 1 is low) | 8 Weeks
  The MAAS (Mindful Attention Awareness Scale) is a 15-item self-report tool that measures an individual's open and receptive awareness of present-moment experiences, with strong psychometric validity and associations with emotional, behavioral, and health outcomes; it can be completed in under 5 minutes, with higher scores indicating greater mindfulness and lower scores reflecting more frequent mind-wandering or inattentiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Reem M Alwhaibi, master, Study Chair — College of Health and Rehabilitation Sciences, Princess Nourah bint Abdulrahman University
Locations (1):
- Cairo University Faculty of Physical Therapy, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
After approval can be shared
Supporting Information: Study Protocol
Time Frame: after 1 month for 12 months
Access Criteria: will upload it to the journal of publication